CLINICAL TRIAL: NCT01548248
Title: An Observational 3-months Study to Evaluate Efficacy and Safety of Insulin Levemir® Used as Basal Insulin on the Glycaemic Control, Weight and Incidence of Hypoglycaemic Events in Insulin Treated Subjects With Type 1 or Type 2 Diabetes
Brief Title: Efficacy and Safety of Levemir® Used as Basal Insulin
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-1928
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; Insulin Aspart

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Levemir® users
  Interventions: Drug: insulin detemir; Drug: insulin aspart

INTERVENTIONS:
Drug: insulin detemir — Prescribed insulin detemir and insulin aspart based on the clinical judgement of the physician. The insulin preparations were prescribed by the physician solely as a result of a normal clinical evaluation. The physician determined the starting dose and frequency, as well as later changes to either dose or frequency, if any.
Drug: insulin aspart — Prescribed insulin detemir and insulin aspart based on the clinical judgement of the physician. The insulin preparations were prescribed by the physician solely as a result of a normal clinical evaluation. The physician determined the starting dose and frequency, as well as later changes to either dose or frequency, if any.

SUMMARY:
This study is conducted in Europe. The aim of this study is to evaluate efficacy and safety of insulin detemir (Levemir®) used as basal insulin on the glycaemic control, weight and incidence of hypoglycaemic events in insulin treated subjects with type 1 or type 2 diabetes treated with insulin NPH under normal clinical practice conditions in Slovakia.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetes treated with insulin NPH

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any subject with type 1 or type 2 diabetes treated with human insulin NPH in whom at the discretion of the participating physicians it was decided to switch insulin treatment to the long-acting insulin analogue insulin detemir in combination with insulin aspart. The selection of the subjects was at the discretion of the participating physicians.
Sampling Method: Non-Probability Sample
Enrollment: 631 (Actual)
Dates: Start 2006-01; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c (glycosylated haemoglobin)

SECONDARY OUTCOMES:
Change in weight
Change in fasting plasma glucose (FPG)
Change in 4-points glucose profiles
Change in lipid profile
Number of hypoglycaemic events
Number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Bratislava, Slovakia

REFERENCES:
- [Result] Zuzana N et al; Effect of Basal Insulin Detemir on Weight and Hypoglycemia in T1DM and T2DM; 2025-PO; 69th Scientific Sessions (2009); American Diabetes Association
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com